CLINICAL TRIAL: NCT06759376
Title: Effects of Vibration Massage and Static Stretching Exercise on Intradialytic Muscle Cramp and Salivary Cortisol Levels: A Randomised Controlled Trial
Brief Title: Vibration Massage, Static Stretching Exercise, Intradialytic Muscle Cramps and Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Figen Akay (Other)
Responsible Party: Sponsor-Investigator, Figen Akay, Specialist Nurse, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-80558721-050.04-240188711
Record Dates: First submitted 2024-12-17; First posted 2025-01-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease; Hemodialysis; Stress
Keywords: Hemodialysis; Stress; intradialytic muscle cramp; Nurse; Vibration Massage; Salivary Cortisol; Static Stretching Exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vibration (Group A) (Experimental): Vibration massage
  Interventions: Other: Vibration massage
- Stretching (Group B) (Experimental): Static stretching exercise
  Interventions: Other: Static stretching exercise
- Control (Group C) (Other): Usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Vibration massage — * Initiation of the stopwatch with the onset of intradialytic muscle cramp,
  * Taking a salivary cortisol test,
  * Performing vibration massage with a vibration massage device for 10 minutes,
  * Visual Analog Scale questioning every 2 minutes during intradialytic muscle cramp,
  * Stopping the stopwatch as soon as the patient states that the intradialytic muscle cramp has ended,
  * Repeat salivary cortisol test at 20 minutes from the onset of intradialytic muscle cramp.
  Arms: Vibration (Group A)
Other: Static stretching exercise — * Initiation of the stopwatch with the onset of intradialytic muscle cramp,
  * Taking a salivary cortisol test,
  * Perform static stretching exercise for 10 minutes,
  * Visual Analog Scale questioning every 2 minutes during intradialytic muscle cramp,
  * Stopping the stopwatch as soon as the patient states that the intradialytic muscle cramp has ended,
  * Repeat salivary cortisol test at 20 minutes from the onset of intradialytic muscle cramp.
  Arms: Stretching (Group B)
Other: Usual Care — * Initiation of the stopwatch with the onset of intradialytic muscle cramp,
  * Taking a salivary cortisol test,
  * Usual care,
  * Visual Analog Scale questioning every 2 minutes during intradialytic muscle cramp,
  * Stopping the stopwatch as soon as the patient states that the intradialytic muscle cramp has ended,
  * Repeat salivary cortisol test at 20 minutes from the onset of intradialytic muscle cramp.
  Arms: Control (Group C)

SUMMARY:
Chronic kidney disease (CKD) is characterised by kidney damage that persists for 3 months or longer or an estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73 m² and is assessed in 6 categories. According to this categorisation, when stage 4 CKD progresses, patients are offered several options for renal replacement therapy. In the last stage of CKD, stage 5, renal replacement therapies including dialysis and kidney transplantation are used. Haemodialysis (HD) is a frequently used life-saving treatment method that removes harmful waste substances accumulated in the body, helps to maintain kidney function, provides fluid-electrolyte balance, prolongs life by managing uremic symptoms. Patients with ESRD are exposed to many health problems such as water-salt balance abnormalities, hypertension, hyperkalemia, metabolic acidosis, hyperphosphatemia, anaemia, cardiovascular disease. While the problems experienced are controlled with HD treatment, the treatment process and the continuation of life dependent on a machine cause life-threatening acute (hypotension, nausea, vomiting, muscle cramps, itching, pain, etc.) and chronic complications (pericarditis, hypertension, anaemia, hepatitis infections, etc.). In addition, due to these complications, HD patients may have problems that cannot be ignored such as deterioration in general health perception, sleep disturbance, anxiety, depression, stress, and difficulties in fulfilling responsibilities due to psychosocial problems. Intradialytic muscle cramp, which develops acutely during HD and is experienced at least once by patients, frequently manifests as involuntary muscle contractions in the lower extremities. The aetiology of intradialytic muscle cramp includes hypotension, electrolyte mineral disorders, high ultrafiltration (UF), excess weight gain between two HDs and carnitine deficiency. In the pharmacological treatment of this complication, which should be managed acutely, intravenous saline solution and hypertonic glucose administration are prominent, but high-quality evidence on the effectiveness of these treatments is needed. While the results of interventions such as aromatherapy, reflexology, massage, stretching-relaxation exercises, hot-cold applications etc. in intradialytic muscle cramp have been reached, the lack of evidence for vibration massage is striking. Management of intradialytic muscle cramp is important for the HD adequacy of patients and failure to manage it may lead to fatal complications such as hypertension, hypervolemia, pulmonary oedema and left ventricular failure due to inadequate HD sessions. It has also been reported that sleep and quality of life are adversely affected in cases where intradialytic muscle cramp cannot be managed; shortening of one HD session per week leads to increased mortality rates, depression and anxiety levels and stress. Salivary cortisol is a useful biomarker often used as a marker of psychological stress. Salivary cortisol levels peak approximately 20 minutes after an acute stress event. Massage, which is among independent nursing interventions, is a manipulation that provides physical and psychological relaxation by mechanically stimulating muscle tissues. During massage, nurses can apply euphlorage, petrissage, friction, tapotman and vibration. Vibration massage is applied to improve muscle atrophy and bone density caused by microgravity and immobilisation. Static stretching exercise, another intervention in intradialytic muscle cramp management, reduces muscle stiffness and tension by increasing muscle flexibility and range of motion by stimulating neural activities. These exercises reduce the risk of injury to joints, muscles and tendons by stimulating the formation of chemicals that allow the connective tissue to move easily and are recommended for the prevention of muscle cramps.

DETAILED DESCRIPTION:
Key words: Vibration massage, Static stretching exercise, Intradialytic muscle cramp, Salivary cortisol level, stress.

Study design: Randomised controlled trial. Objectives:The aim of this randomised controlled clinical trial was to evaluate the effect of vibration massage and static stretching exercise on intradialytic muscle cramp (severity and duration) and salivary cortisol levels during intradialytic muscle cramp.

Phase of the study: For this study, permission was obtained from Eskişehir Osmangazi University Clinical Research Ethics Committee that there was no ethical objection. For the financial support of the study, an application was made to the Scientific and Technological Research Council of Türkiye (TUBITAK), a state institution in Turkey, and the result is awaited. After approval, the data collection phase will begin.

Interventional Study Model: Factorial Vibration massage group (Group A), Static stretching exercise (Group B), Control Group (Group C).

Masking: Outcomes Assessor. Allocation: Stratified Randomized. Enrollment: The total number of participants to be enrolled in the clinical study was determined as 30.

Biospecimen Retention: Collection of saliva for salivary cortisol testing at the time of intradialytic muscle cramp and at 20 minutes after the patients to be included in the study.

Target Follow-Up Duration: Participants will be followed up at the time of intradialytic muscle cramp and at the time of its termination.

Intervention First intervention group: Vibration massage (Group A).

* Initiation of the stopwatch with the onset of intradialytic muscle cramp,
* Taking a salivary cortisol test,
* 10 minutes of vibration massage,
* VAS questioning every 2 minutes during intradialytic muscle cramp,
* Stopping the stopwatch as soon as the patient states that the intradialytic muscle cramp has ended,
* Repeat salivary cortisol test at 20 minutes from the onset of intradialytic muscle cramp.

The second group of intervention: Static stretching exercise (Group B)

* Initiation of the stopwatch with the onset of intradialytic muscle cramp,
* Taking a salivary cortisol test,
* Perform static stretching exercise for 10 minutes,
* VAS questioning every 2 minutes during intradialytic muscle cramp,
* Stopping the stopwatch as soon as the patient states that the intradialytic muscle cramp has ended,
* Repeat salivary cortisol test at 20 minutes from the onset of intradialytic muscle cramp.

Control group: Usual care (Group C)

* Initiation of the stopwatch with the onset of intradialytic muscle cramp,
* Taking a salivary cortisol test,
* Usual care,
* VAS questioning every 2 minutes during intradialytic muscle cramp,
* Stopping the stopwatch as soon as the patient states that the intradialytic muscle cramp has ended,
* Repeat salivary cortisol test at 20 minutes from the onset of intradialytic muscle cramp.

Outcome Measures

Primary Outcome Measure Information:

* The effect of vibration massage on the severity, duration and salivary cortisol level of intradialytic muscle cramp.
* The effect of static stretching exercise on intradialytic muscle cramp severity, duration and salivary cortisol level.
* To determine which intervention (vibration massage and static stretching exercise) is more effective on intradialytic muscle cramp severity, duration and salivary cortisol level.

Secondary Outcome Measure: The effectiveness of vibration massage and stretching exercise interventions for acute stress management will be determined.

Age Limits: Patients aged 18 years and older. Eligibility Criteria: 18 years of age and over, conscious, Turkish speaking and understanding, accepting the research, With a normal body mass index (18.5-24.9), Patients with intradialytic muscle cramps in the lower limb.

Statistical Analysis Plan: The data obtained in the study will be analysed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 programme. The statistician performing the statistics of the data will not be informed which group the patients are in and the interventions applied to the groups, thus statistical blinding will be ensured. Kolmogorov Smirnov Test will be used to determine whether the research data are normally distributed. According to the Kolmogorov Smirnov Test, if p>0.05, it is determined that the distribution is normal. However, if p<0.05, it is determined that the distribution is not normal and the Skewness and Kurtosis values of the data are examined. If Skewness and Kurtosis values are between +2 and -2, it is accepted that the variable shows normal distribution. Homogeneity of descriptive characteristics between groups will be tested by chi-square analysis. For the difference between group averages, one-way analysis of variance will be used if the data are normally distributed, and Kruskal Wallis test will be used if the data are not normally distributed. Changes in measurements within the group will be analysed by repeated measures ANOVA test if the data are normally distributed, and by Friedman test if the data are not normally distributed.

Informed Consent Form: Informed Voluntary Consent signature will be obtained from patients who agree to participate in the study. The research will be conducted in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over, conscious, Turkish speaking and understanding, accepting the research,
* Patients with normal body mass index (18.5-24.9) [Since body mass can affect the distribution of vibration and cortisol level, it was planned to include patients with normal body mass index in the sample].
* Patients with intradialytic muscle cramp in the lower extremities will be included [Although intradialytic cramp often occurs in the lower extremities, vibration massage and static stretching exercise will be applied to the same muscle group (gastrocnemius and soleus muscles) in the lower extremities to keep the variables under control].

Exclusion Criteria:

* Intradialytic muscle cramps in the upper extremity,
* Intradialytic muscle cramps, those with incomplete tissue integrity in the region and thrombophlebitis, hematoma, etc. [In order for vibration massage to be performed, individuals must have skin integrity and normal blood characteristics.]
* Those with foot deformation,
* Those who use anti-inflammatory, analgesic drugs and those who additionally use adjuvant therapy (antidepressants, anticonvulsants, muscle relaxants, etc.) up to 4 hours before the HD session, as intradialytic muscle cramps and their duration may be affected,
* Those who are taking routine cortisone treatment and medications with hormonal effects (oral contraceptives, steroid-containing bronchodilators, etc.) so that the salivary cortisol test is not affected.

  --Alcohol users,
* Hypoglycemic patients,
* Patients with psychiatric diagnosis and those using medication related to this diagnosis,
* Patients with mouth ulcers, inflammation, etc.
* Patients who ate or drank anything other than water, chewed gum, or consumed foods or beverages containing citric acid 15 minutes before intradialytic muscle cramping,
* Patients who use high doses of biotin (>5 mg/day) and whose last biotin treatment has not passed 8 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
intradialytic muscle cramp (severity) | 1 year
  * Visual Analog Scale questioning will be performed every 2 minutes during the intradialytic cramp period.
  * The effect of 10 minutes of vibration massage and static stretching exercise interventions on the severity of intradialytic muscle cramp will be examined.
Salivary cortisol levels | 1 year
  * The stress level of the patient during intradialytic muscle cramp will be quantitatively assessed by salivary cortisol testing.
  * Salivary cortisol tests will be taken again at 20 minutes to evaluate the effectiveness of vibration massage and static stretching exercise interventions applied to intradialytic muscle cramp for 10 minutes and to evaluate which intervention is superior.
  * The effect of vibration massage and static stretching exercise on salivary cortisol level will be evaluated.
intradialytic muscle cramp (duration) | 1 year
  * Intradialytic muscle cramp duration will be measured with a stopwatch.
  * The effect of 10 minutes of vibration massage and static stretching exercise interventions on muscle cramp duration will be examined.

SECONDARY OUTCOMES:
Acute stress | 1 year
  -In acute stress management, the effectiveness of the interventions will be evaluated by applying 10 minutes of vibration massage to 10 hemodialysis patients, 10 minutes of static stretching exercise to 10 hemodialysis patients, and usual care to 10 hemodialysis patients, with a salivary cortisol test taken at the 20th minute.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Özkaraman, Professor, Study Director — Eskisehir Osmangazi University Faculty of Health Sciences
Locations (1):
- Private Anatolian Dialysis Center, Eskişehir, Turkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Summary data can be provided starting 6 months after publication.
Supporting Information: Study Protocol, SAP
Time Frame: July - December 2025
Access Criteria: Academic staff can request this information. Data can be shared with the permission of all researchers involved in the study.

REFERENCES:
- [Background] Zoccali C, Mallamaci F, Adamczak M, de Oliveira RB, Massy ZA, Sarafidis P, Agarwal R, Mark PB, Kotanko P, Ferro CJ, Wanner C, Burnier M, Vanholder R, Wiecek A. Cardiovascular complications in chronic kidney disease: a review from the European Renal and Cardiovascular Medicine Working Group of the European Renal Association. Cardiovasc Res. 2023 Sep 5;119(11):2017-2032. doi: 10.1093/cvr/cvad083. PMID 37249051
- [Background] Youdas JW, Krause DA, Egan KS, Therneau TM, Laskowski ER. The effect of static stretching of the calf muscle-tendon unit on active ankle dorsiflexion range of motion. J Orthop Sports Phys Ther. 2003 Jul;33(7):408-17. doi: 10.2519/jospt.2003.33.7.408. PMID 12918866
- [Background] Yilmaz Menek M, Dansuk E, Tayboga UI. Effect of Local Vibration Therapy on Pain, Joint Position Sense, Kinesiophobia, and Disability in Cervical Disc Herniation: A Randomized Controlled Trial. J Clin Med. 2024 Aug 5;13(15):4566. doi: 10.3390/jcm13154566. PMID 39124832
- [Background] Trajano GS, Taylor JL, Orssatto LBR, McNulty CR, Blazevich AJ. Passive muscle stretching reduces estimates of persistent inward current strength in soleus motor units. J Exp Biol. 2020 Nov 5;223(Pt 21):jeb229922. doi: 10.1242/jeb.229922. PMID 32978317
- [Background] Skrinjar I, Loncar Brzak B, Vidranski V, Vucicevic Boras V, Rogulj AA, Pavelic B. Salivary Cortisol Levels and Burning Symptoms in Patients with Burning Mouth Syndrome before and after Low Level Laser Therapy: a Double Blind Controlled Randomized Clinical Trial. Acta Stomatol Croat. 2020 Mar;54(1):44-50. doi: 10.15644/asc54/1/5. PMID 32523156
- [Background] Suleymanlar G, Utas C, Arinsoy T, Ates K, Altun B, Altiparmak MR, Ecder T, Yilmaz ME, Camsari T, Basci A, Odabas AR, Serdengecti K. A population-based survey of Chronic REnal Disease In Turkey--the CREDIT study. Nephrol Dial Transplant. 2011 Jun;26(6):1862-71. doi: 10.1093/ndt/gfq656. Epub 2010 Nov 4. PMID 21051501
- [Background] Needs D, Blotter J, Cowan M, Fellingham G, Johnson AW, Feland JB. Effect of Localized Vibration Massage on Popliteal Blood Flow. J Clin Med. 2023 Mar 4;12(5):2047. doi: 10.3390/jcm12052047. PMID 36902835
- [Background] Mastnardo D, Lewis JM, Hall K, Sullivan CM, Cain K, Theurer J, Huml A, Sehgal AR. Intradialytic Massage for Leg Cramps Among Hemodialysis Patients: a Pilot Randomized Controlled Trial. Int J Ther Massage Bodywork. 2016 Jun 3;9(2):3-8. doi: 10.3822/ijtmb.v9i2.305. eCollection 2016 Jun. PMID 27257445
- [Background] Mantilla-Manosalva N, Guadarrama S, Bedoya-Munoz LJ, Giraldo-Moreno S, Cuellar-Valencia L, Iriarte-Aristizabal MF, Leon MX, Mendoza-Montenegro FA, Correa-Morales JE. Pharmacological Treatment for Dialysis-Related Muscle Cramps: A Systematic Review. Semin Dial. 2024 Nov-Oct;37(6):415-423. doi: 10.1111/sdi.13223. Epub 2024 Aug 18. PMID 39155056
- [Background] Lupowitz L. Vibration Therapy - A Clinical Commentary. Int J Sports Phys Ther. 2022 Aug 1;17(6):984-987. doi: 10.26603/001c.36964. eCollection 2022. No abstract available. PMID 36237646
- [Background] Lee DY, Kim E, Choi MH. Technical and clinical aspects of cortisol as a biochemical marker of chronic stress. BMB Rep. 2015 Apr;48(4):209-16. doi: 10.5483/bmbrep.2015.48.4.275. PMID 25560699
- [Background] Imai T, Nagamatsu T, Yoshizato Y, Miyara K, Sumizono M, Nakamura M. Acute Effects of Handheld Vibration Massage on Posterior Shoulder Soft Tissues. Int J Sports Phys Ther. 2024 Aug 2;19(8):1003-1011. doi: 10.26603/001c.121299. eCollection 2024. PMID 39100939
- [Background] Hill NR, Fatoba ST, Oke JL, Hirst JA, O'Callaghan CA, Lasserson DS, Hobbs FD. Global Prevalence of Chronic Kidney Disease - A Systematic Review and Meta-Analysis. PLoS One. 2016 Jul 6;11(7):e0158765. doi: 10.1371/journal.pone.0158765. eCollection 2016. PMID 27383068
- [Background] Higaki Y, Yamato Y, Fujie S, Inoue K, Shimomura M, Kato S, Horii N, Ogoh S, Iemitsu M. Acute effects of the different relaxation periods during passive intermittent static stretching on arterial stiffness. PLoS One. 2021 Nov 15;16(11):e0259444. doi: 10.1371/journal.pone.0259444. eCollection 2021. PMID 34780500
- [Background] Heo EH, Kim S, Park HJ, Kil SY. The effects of a simulated laughter programme on mood, cortisol levels, and health-related quality of life among haemodialysis patients. Complement Ther Clin Pract. 2016 Nov;25:1-7. doi: 10.1016/j.ctcp.2016.07.001. Epub 2016 Jul 27. PMID 27863598
- [Background] Hao G, Lu W, Huang J, Ding W, Wang P, Wang L, Ding F, Hu M, Hou L. Predialysis fluid overload linked with quality of sleep in patients undergoing hemodialysis. Sleep Med. 2018 Nov;51:140-147. doi: 10.1016/j.sleep.2018.07.011. Epub 2018 Jul 31. PMID 30165338
- [Background] Hassanzadeh M, Kiani F, Bouya S, Zarei M. Comparing the effects of relaxation technique and inhalation aromatherapy on fatigue in patients undergoing hemodialysis. Complement Ther Clin Pract. 2018 May;31:210-214. doi: 10.1016/j.ctcp.2018.02.019. Epub 2018 Mar 6. PMID 29705457
- [Background] Hargrove N, El Tobgy N, Zhou O, Pinder M, Plant B, Askin N, Bieber L, Collister D, Whitlock R, Tangri N, Bohm C. Effect of Aerobic Exercise on Dialysis-Related Symptoms in Individuals Undergoing Maintenance Hemodialysis: A Systematic Review and Meta-Analysis of Clinical Trials. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):560-574. doi: 10.2215/CJN.15080920. Epub 2021 Mar 25. PMID 33766925
- [Background] Hammerfald K, Eberle C, Grau M, Kinsperger A, Zimmermann A, Ehlert U, Gaab J. Persistent effects of cognitive-behavioral stress management on cortisol responses to acute stress in healthy subjects--a randomized controlled trial. Psychoneuroendocrinology. 2006 Apr;31(3):333-9. doi: 10.1016/j.psyneuen.2005.08.007. Epub 2005 Sep 23. PMID 16183205
- [Background] Frisch JU, Hausser JA, Mojzisch A. The Trier Social Stress Test as a paradigm to study how people respond to threat in social interactions. Front Psychol. 2015 Feb 2;6:14. doi: 10.3389/fpsyg.2015.00014. eCollection 2015. PMID 25698987
- [Background] Flythe JE, Hilliard T, Castillo G, Ikeler K, Orazi J, Abdel-Rahman E, Pai AB, Rivara MB, St Peter WL, Weisbord SD, Wilkie C, Mehrotra R. Symptom Prioritization among Adults Receiving In-Center Hemodialysis: A Mixed Methods Study. Clin J Am Soc Nephrol. 2018 May 7;13(5):735-745. doi: 10.2215/CJN.10850917. Epub 2018 Mar 20. PMID 29559445
- [Background] Fujiwara K, Asai H, Toyama H, Kunita K, Yaguchi C, Kiyota N, Tomita H, Jacobs JV. Changes in muscle thickness of gastrocnemius and soleus associated with age and sex. Aging Clin Exp Res. 2010 Feb;22(1):24-30. doi: 10.1007/BF03324811. Epub 2009 Nov 6. PMID 19920407
- [Background] Dickmeis T. Glucocorticoids and the circadian clock. J Endocrinol. 2009 Jan;200(1):3-22. doi: 10.1677/JOE-08-0415. Epub 2008 Oct 29. PMID 18971218
- [Background] Bruck K, Stel VS, Gambaro G, Hallan S, Volzke H, Arnlov J, Kastarinen M, Guessous I, Vinhas J, Stengel B, Brenner H, Chudek J, Romundstad S, Tomson C, Gonzalez AO, Bello AK, Ferrieres J, Palmieri L, Browne G, Capuano V, Van Biesen W, Zoccali C, Gansevoort R, Navis G, Rothenbacher D, Ferraro PM, Nitsch D, Wanner C, Jager KJ; European CKD Burden Consortium. CKD Prevalence Varies across the European General Population. J Am Soc Nephrol. 2016 Jul;27(7):2135-47. doi: 10.1681/ASN.2015050542. Epub 2015 Dec 23. PMID 26701975
- [Background] Blair J, Adaway J, Keevil B, Ross R. Salivary cortisol and cortisone in the clinical setting. Curr Opin Endocrinol Diabetes Obes. 2017 Jun;24(3):161-168. doi: 10.1097/MED.0000000000000328. PMID 28375882
- [Background] Atkinson AJ Jr. Elucidation of the pathophysiology of intradialytic muscle cramps: pharmacokinetics applied to translational research. Transl Clin Pharmacol. 2019 Dec;27(4):119-122. doi: 10.12793/tcp.2019.27.4.119. Epub 2019 Dec 31. PMID 32095478
- [Background] Alghadir AH, Anwer S, Zafar H, Iqbal ZA. Effect of localised vibration on muscle strength in healthy adults: a systematic review. Physiotherapy. 2018 Mar;104(1):18-24. doi: 10.1016/j.physio.2017.06.006. Epub 2017 Aug 6. PMID 28947078
- [Background] Ahsan M, Gupta M, Omar I, Frinak S, Gendjar S, Osman-Malik Y, Yee J. Prevention of hemodialysis-related muscle cramps by intradialytic use of sequential compression devices: a report of four cases. Hemodial Int. 2004 Jul 1;8(3):283-6. doi: 10.1111/j.1492-7535.2004.01106.x. PMID 19379428